CLINICAL TRIAL: NCT02878408
Title: Immuno-Génétique, Inflammation, Retro-Virus, Environnement
Brief Title: Immuno-Genetic, Inflammation, Retro-Virus, Environment
Acronym: I-Give
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pr. Marion Leboyer (Other)
Collaborators: National Research Agency, France (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor-Investigator, Pr. Marion Leboyer, Responsible for Pôle de psychiatrie of Hospital Albert Chenevier- Henri Mondor, Fondation FondaMental
Organization: Fondation FondaMental (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: I-Give; IDRCB : 2013-A01639-36 (Other: ANSM)
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Bipolar Disorder; Schizophrenia
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- acute Bipolar disorder (Other): blood sampling and data collection Following visit at end of hospitalisation (blood sampling and data collection)
  Interventions: Genetic: Blood sampling
- acute Schizophrenia (Other): blood sampling and data collection Following visit at end of hospitalisation (blood sampling and data collection)
  Interventions: Genetic: Blood sampling
- stable Bipolar disorder (Other): blood sampling and data collection (only one visit)
  Interventions: Genetic: Blood sampling
- stable Schizophrenia (Other): blood sampling and data collection (only one visit)
  Interventions: Genetic: Blood sampling
- healthy control (Other): blood sampling and data collection (only one visit)
  Interventions: Genetic: Blood sampling
- TOC (Other): blood sampling and data collection (only one visit)
  Interventions: Genetic: Blood sampling

INTERVENTIONS:
Genetic: Blood sampling — supplementary blood sampling for analysis of: immuno-genetic, inflammatory process, retro-viruses activity, Questionaries about environment risk factors

SUMMARY:
Immunology combined to neurobiology now offer prominent tools to yield biomarkers, so far missing in psychiatry, and to design innovative treatment approaches based on the discovery of new molecular and cellular targets. As Bipolar Disorder and Schizophrenia are now known to be significantly associated with neuro-inflammation, the project I-GIVE will combine multidisciplinary approaches (clinical, viral, immunological, genetic) to explore a global hypothesis placing the Human Endogenous Retro-Virus, HERV-W, at the crossroads between susceptibility to environmental factors (such as winter-spring births, infections, urbanicity…) and genetic factors controlling immune responses.

Thus I-GIVE will allow identification of new biomarkers and their correlation with clinical profiles and immuno-inflammatory/immuno-genetic markers, and description of patho-physiological mechanisms of a psychiatric disorder. In addition, I-GIVE should help to design innovative treatments and foster personalized psychiatry tailored to the needs of each patient. Notably, monoclonal antibodies anti-HERV-W Env will be assessed in a preclinical model for their ability to slow, stop, or even reverse the progression of the psychosis in patients. I-GIVE project should thus lead to major results that will have strong impacts on the scientific community, pharmaceutical industries and, in a longer term, on improvement of patients suffering Bipolar Disorder or Schizophrenia and their family.

DETAILED DESCRIPTION:
The investigators and others have been able to demonstrate that HERV-W envelope gene (Env) encodes a pro-inflammatory and neurotoxic protein after reactivation by environmental factors. In this context, the investigators have reported preliminary data showing an association between Human Endogenous Retroviruses type "W" family (HERV-W) and major psychotic disorder, bipolar disorder (BD) and schizophrenia (SZ) : In 2008, the investigators reported for the first time, the presence of ENV protein in the serum of 50 % of SZ patients associated with a chronic inflammatory status reflected by elevated serum level of C-Reactive Protein (CRP). The investigators have been able to confirm this finding and extend it to BD and showed an elevation of HERV-W RNA transcripts both in BD and SZ as compared to healthy controls. Furthermore, the investigators also observed for the first time that toxoplasma Gondii, known to be able to induce reactivation of HERV-W, is associated with an increased risk to develop BD (OR: 2.3) close to the one previously observed in SZ (OR= 2.17)

The present project I-GIVE aims to extend and refine such findings and to obtain a proof of concept of the involvement of Human Endogenous Retrovirus elements in bipolar disorder and schizophrenia. I-GIVE is divided into four complementary scientific tasks:

1. assessing the systemic HERV-W (ENV and GAG) antigen serum levels and the RNA and DNA copy number variants of stabilized and acutely ill patients,
2. measuring the systemic associated immuno-inflammatory cascade in BD patients at different stages of the disorder and occurrence of medical comorbidities,
3. identifying the clinical characteristics of patients according to HERV-W expression and immuno-inflammatory profiles,
4. exploring the gene (immuno-genetic) x environment interactions that may modulate the immuno-inflammatory response

Clinical and biological data from acute BP and SZ patients will be compared first with themselves at two different times. They will be compared also to healthy control's data, and third to stabilised BP and SZ patients.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar disorder or Schizophrenia (according to Diagnostic and Statistical Manual of Mental Disorders IV)

Exclusion Criteria:

* pregnant women
* Vaccination within 4 precedent weeks
* Severe neurologic illness
* Immunosuppressing or immuno-modulating treatment.
* Infectious disease within 4 precedent weeks (including HIV 1 et 2, Hepatite B, C)
* Refuse to have HIV and hepatite B et C tests or to be informed of their results

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2014-11; Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
HERV-W | inclusion
  measure of HERV retroviral DNA, RNA and envelop proteins

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Psychiatry Department of Perrens Hospital, Bordeaux
  - Clinical Investigations Center of Mondor Hospital, Créteil
  - Psychiatry Department of Mondor Hospital, Créteil
  - Psychiatry Department of Widal Hospital, Paris
  - EPS Maison Blanche, Paris
  - Psychiatry Department of R. Dubos Hospital, Pontoise

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.fondation-fondamental.org/